CLINICAL TRIAL: NCT02086110
Title: A Pilot Study Examining Microbiota Composition in Children With Autism and Gastrointestinal Symptoms After Use of Bifidobacterium Infantis and Milk Oligosaccharides
Brief Title: Effect of Milk Oligosaccharides and Bifidobacteria on the Intestinal Microflora of Children With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 450072
Record Dates: First submitted 2014-03-07; First posted 2014-03-13 (Estimated); Results first posted 2019-08-01 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-05

CONDITIONS: Autism
Keywords: probiotic; prebiotic; autism; oligosaccharides; Bifidobacterium infantis
MeSH Terms: conditions — Autistic Disorder | interventions — Synbiotics; Prebiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prebiotic only first, then synbiotic (Active Comparator): This group will receive prebiotic only (bovine milk oligosaccharides, administered orally twice per day for a daily total of 0.3 g per pound of body weight) for the first five weeks, followed by a two week break with no treatment, and then will receive the synbiotic (Bifidobacterium infantis (10 billion CFU) twice a day plus 0.3 g per pound body weight of bovine milk oligosaccharides in two divided doses per day orally) for the next five weeks.
  Interventions: Dietary Supplement: Synbiotic; Dietary Supplement: Prebiotic
- Synbiotic first, then prebiotic only (Active Comparator): This group will receive the synbiotic (Bifidobacterium infantis (10 billion CFU) twice a day plus 0.3 g per pound body weight of bovine milk oligosaccharides in two divided doses per day orally) for the first five weeks, followed by a two week break with no treatment, and then will receive the prebiotic only (bovine milk oligosacharrides, administered orally twice per day for a daily total of 0.3 g per pound of body weight) for the next five weeks.
  Interventions: Dietary Supplement: Synbiotic; Dietary Supplement: Prebiotic

INTERVENTIONS:
Dietary Supplement: Synbiotic
  Other Names: Bifidobacterium infantis SC268; bovine colostrum, bovine oligosaccharides
Dietary Supplement: Prebiotic
  Other Names: bovine colostrum, bovine oligosaccharides

SUMMARY:
The purpose of this study is to determine the tolerability of dietary supplements and if these supplements can promote a healthy bacterial environment in the intestines of children with autism spectrum disorders and gastrointestinal complaints.

DETAILED DESCRIPTION:
This study investigates the feasibility, tolerability, and effects of a dietary supplement on the intestinal flora of children with autism spectrum disorders. This study is divided into two parts, each five weeks long, with a two week break in between. During one part of the study, a prebiotic (milk oligosaccharides from bovine colostrum) will be given. During the other part of the study, the synbiotic composed of the prebiotic and probiotic (bifidobacterium infantis) will be given. Stool will be analyzed at the end of each study arm to determine content of bifidobacteria.

On May 8, 2018, we updated the study start and completion dates to the actual (instead of anticipated) dates.

On May 30-31, 2019, we updated the study results section.

ELIGIBILITY:
Inclusion Criteria:

* Autism
* Diarrhea and/or constipation

Exclusion Criteria:

* Milk protein or other documented food allergy
* Lactose intolerance
* Compromised Immunity
* GI conditions (inflammatory bowel disease, celiac disease, short gut, etc.)
* Systemic steroid, antifungal, or antibiotic use within a month of starting the study
* Failure to thrive
* Medically prescribed diets or supplements (including probiotic use within the past month).
* Vegetarian or dairy restricted diet
* Other medical conditions (seizures, genetic disorders, liver/pancreatic disease, cystic fibrosis, etc.)
* Medications that interfere or alter intestinal motility or microbiota composition.
* Full scale intelligence quotient (IQ) <40

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2014-06-06 (Actual); Primary Completion 2015-11-16 (Actual); Study Completion 2015-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Angkustsiri, MD, Principal Investigator — UC Davis MIND Institute
Locations (1):
- UC Davis MIND Institute, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prebiotic Only First, Then Synbiotic | Synbiotic First, Then Prebiotic Only
Started | 5 | 6
Completed | 4 | 5
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prebiotic Only First, Then Synbiotic | Synbiotic First, Then Prebiotic Only | Total
Number analyzed (Participants) | 5 | 6 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 6 | 11
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 4 | 5 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, non-Hispanic | 3 | 5 | 8
  African-American, non-Hispanic | 1 | 0 | 1
  White, Hispanic/Latino | 1 | 1 | 2
  African-American, Hispanic/Latino | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Stool Microbiota Composition Change During Prebiotic Only Treatment
Description: The stool microbiome composition will be analyzed through next generation sequencing and quantitative polymerase chain reaction. Overall bacterial composition change is reported here, as change in enterotype from before prebiotic only treatment to after prebiotic treatment, for all subjects. Enterotypes were organized into four categories for analysis: a community high in Prevotella ("Prevotella"), a community high in Bifidobacterium ("Bifidobacterium"), a community high in Bacteroides ("Bacteroides"), and a mixed community ("Mixed") that did not fall into one of the other three enterotypes but instead consisted of a varied combination of bacteria, including among others Akkermansia, Collinsela, Prevotella, and/or Bacteroides.
Time Frame: Five weeks
Population: In the Prebiotic First group, 1 subject withdrew consent prior to providing stool sample. In the Synbiotic First group, 1 subject withdrew consent prior to starting prebiotic treatment, and 1 subject was unable to provide a stool sample for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Prebiotic Only First, Then Synbiotic | Synbiotic First, Then Prebiotic Only
Number analyzed (Participants) | 4 | 4
Participants
  No change in enterotype | 2 | 3
  Bifidobacterium to Prevotella | 1 | 0
  Bacteroides to Bifidobacterium | 1 | 0
  Prevotella to Bifidobacterium | 0 | 1

2. Primary Outcome: Stool Microbiota Composition Change During Synbiotic Treatment
Description: The stool microbiome composition will be analyzed through next generation sequencing and quantitative polymerase chain reaction. Overall bacterial composition change is reported here, as change in enterotype from before synbiotic treatment to after synbiotic treatment, for all subjects. Enterotypes were organized into four categories for analysis: a community high in Prevotella ("Prevotella"), a community high in Bifidobacterium ("Bifidobacterium"), a community high in Bacteroides ("Bacteroides"), and a mixed community ("Mixed") that did not fall into one of the other three enterotypes but instead consisted of a varied combination of bacteria, including among others Akkermansia, Collinsela, Prevotella, and/or Bacteroides.
Time Frame: Five weeks
Population: In the Prebiotic First group, 1 subject withdrew consent prior to starting synbiotic treatment. In the Synbiotic First group, 1 subject withdrew consent prior to providing stool sample, and 1 subject was unable to provide a stool sample for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Prebiotic Only First, Then Synbiotic | Synbiotic First, Then Prebiotic Only
Number analyzed (Participants) | 4 | 4
Participants
  No change in enterotype | 4 | 2
  Prevotella to Mixed | 0 | 1
  Prevotella to Bifidobacterium | 0 | 1

3. Secondary Outcome: Serum Immune Profile Change During Prebiotic Only Treatment
Description: Luminex technology will be used to determine a serum immune profile of each participants in response to the study supplement. This profile included assessment of change in percentage of stimulated CD4+ T cells producing intracellular IL-13 before and after Synbiotic treatment ("Post-Synbiotic % IL-13"), and assessment of change in percentage of stimulated CD8+ T cells producing TNF-alpha before and after Prebiotic Only treatment ("Post-Prebiotic % TNF-alpha"). Results are reported here for all subjects regardless of treatment order assignment. Decrease in inflammatory cytokines IL-13 and TNF-alpha is interpreted as a positive outcome.
Time Frame: Five weeks
Population: 1 subject was unable to provide blood specimens throughout the study due to significant anxiety with regard to venipuncture, so only 7 subjects' serum was available for analysis.
Measure: Median (95% Confidence Interval); unit: percentage of cytokine production
Groups:
- All Subjects: All subjects with serum samples available for analysis were included below.
Arm/Group | All Subjects
Number analyzed (Participants) | 7
percentage of cytokine production
  Post-Synbiotic % IL-13 | -0.8 [-2.073 to -0.524]
  Post-Prebiotic % TNF-alpha | -7.9 [-14.375 to -1.425]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from time of consent through end-of-treatment (12 weeks total).
Groups:
- Prebiotic Only Arm: Includes reported adverse events for all subjects while receiving prebiotic only (bovine milk oligosaccharides, administered orally twice per day for a daily total of 0.3 g per pound of body weight).
- Synbiotic Arm: Includes reported adverse events for all subjects while receiving the synbiotic (Bifidobacterium infantis (10 billion CFU) twice a day plus 0.3 g per pound body weight of bovine milk oligosaccharides in two divided doses per day orally).
Arm/Group | Prebiotic Only Arm | Synbiotic Arm
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 10/10 | 10/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prebiotic Only Arm (N=10) | Synbiotic Arm (N=10)
Increased gassiness (Gastrointestinal disorders) | 2 (2) | 2 (2)
Stomachache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Sleep disturbances (Psychiatric disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (4) | 2 (4)
Constipation (Gastrointestinal disorders) | 2 (4) | 2 (4)
Pain associated with bowel movements (Gastrointestinal disorders) | 3 (3) | 3 (3)
Bloating (Gastrointestinal disorders) | 1 (1) | 2 (2)
Lethargy (Psychiatric disorders) | 1 (1) | 0 (0)
Weight gain (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hives (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Lack of a clear control group receiving a placebo, resulting in possible placebo effect (partially addressed by study's cross-over design). Study duration was short. Lack of a probiotic only arm to parse out specific treatment effects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes